CLINICAL TRIAL: NCT00548600
Title: A Randomized Clinical Trial Comparing Radical Radiotherapy by External Beam Radiation Versus Radical Radiotherapy Using a Combination of a Temporaory Iridium Implant Plus External Beam Radiation in Surgically Staged B2 and C Carcinoma of the Prostate
Brief Title: Radical Radiotherapy by External Beam Radiation Versus Radical Radiotherapy With Temporary Iridium Implant Plus External Beam Radiation in Carcinoma of the Prostate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-1992-Iridium
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Last update posted 2007-10-24 (Estimated); Status verified 2007-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Iridium; Implant; Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Iridium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Iridium implant plus external beam irradiation
  Interventions: Procedure: Iridium Implant
- 2 (Active Comparator): Standard external beam irradiation alone
  Interventions: Radiation: Standard external beam irradiation

INTERVENTIONS:
Procedure: Iridium Implant — Temporary iridium implant of the prostate will be done and a dose of 3000 cGy will be delivered in the next 48-72 hours. Two weeks later 20 fractions of external beam radiation at a dose of 4000 cGy will be administered over a period of 4 weeks.
  Arms: 1
Radiation: Standard external beam irradiation — Standard external beam irradiation at a dose of 6400 cGy in 32 fractions over 6 and a half weeks will be administered.
  Arms: 2

SUMMARY:
The specific objective of this study is to compare the relative efficacy of the combination of a temporary iridium implant plus external beam irradiation versus standard external beam irradiation alone in patients with Stage B2 and C prostatic carcinoma. Benefit will be assessed in terms of local recurrence, survival, and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically proven adenocarcinoma of the prostate
* The primary tumour should be staged clinically B2 or C as classified by A.J.C. Staging System

Exclusion Criteria:

* Patients requiring transurethral prostatectomy (TURP) prior to diagnosis
* Presence of metastases identified by bone scan, chest x-ray or CT scan of the abdomen and pelvis, or staging lymphadenectomy
* Karnofsky performance status less than 80
* Inadequate laboratory results: i.e. Hb < 12 gm/litre, WBC < 3.5 x 10 per litre, platelets < 100 x 10/litre, urea > 13 mmol/litre, creatinine > 220 mmol/litre
* Unfit for surgery for other medical reasons
* Age above 75 years
* Failure to provide written informed consent

Max Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 1992-05; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Rate of local control as determined by biopsy at 18 months | 18-months

SECONDARY OUTCOMES:
Distant metastasis | survival
Overall mortality | survival
Mortality due to prostate cancer | survival
Local complications of radiation | 2-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jinka Sathya, MD, Study Chair — Juravinski Cancer Centre
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Sathya JR, Davis IR, Julian JA, Guo Q, Daya D, Dayes IS, Lukka HR, Levine M. Randomized trial comparing iridium implant plus external-beam radiation therapy with external-beam radiation therapy alone in node-negative locally advanced cancer of the prostate. J Clin Oncol. 2005 Feb 20;23(6):1192-9. doi: 10.1200/JCO.2005.06.154. PMID 15718316